CLINICAL TRIAL: NCT02185482
Title: Physician Led Counseling for Depression in Type 2 Diabetes Mellitus: A Randomized, Controlled Trial
Brief Title: Physician Led Counseling in Management of Depression in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adwin Life Care (Industry)
Collaborators: NMP Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Adwin112
Record Dates: First submitted 2014-07-04; First posted 2014-07-09 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Depression; Type 2 Diabetes Mellitus
Keywords: Psychological counselling; Randomized single blind study; Depression; Diabetes
MeSH Terms: conditions — Depression; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physician Supported Care (Experimental): The intervention is an individualized, stepped-care depression treatment program provided by a depression clinical specialist primary care physician.
  Interventions: Behavioral: Physician Supported Care
- Usual care (Other): Usual care patients will be advised to consult with their primary care physician regarding depression. Primary care physicians prescribe antidepressant medication and can refer patients to the Mental Health Services.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Physician Supported Care
  Arms: Physician Supported Care
Other: Usual care
  Arms: Usual care

SUMMARY:
There is a high prevalence of depression in patients with diabetes mellitus. Depression has been shown to be associated with poor self-management (adherence to diet, exercise, checking blood glucose levels) levels in patients with diabetes.To determine whether enhancing quality physician's care for depression improves both depression and diabetes outcomes in patients with depression and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are ambulatory,
* Had adequate hearing to complete a telephone interview,
* Diabetic patients screened for depression

Exclusion Criteria:

* Currently in care with a psychiatrist;
* Diagnosis of bipolar disorder or schizophrenia;
* Use of antipsychotic or mood stabilizer medication
* Mental confusion on interview, suggesting significant dementia.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
change in depression using SCL-90 depression scale | Change from baseline to six month

SECONDARY OUTCOMES:
Glycemic control measured using glycosylated hemoglobin levels | Change from baseline to six month

OTHER OUTCOMES:
Global assessment of improvement using Patient Global Impression | Change from baseline to six months

CONTACTS AND LOCATIONS:
Overall Officials: Ram Sharma, MD, Study Director — NMP Medical Research Institute; Naresh C Kumar, MD, Principal Investigator — Kaithal Civil Hospital
Locations (2):
- India (2):
  - NMP Medical Research Institute, Kaithal, Haryana
  - GyanSanjeevani, Jaipur, Rajasthan